CLINICAL TRIAL: NCT06877650
Title: A Phase 1 Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Preliminary Anti-tumor Activity of JMT108 Injection in Participants With Advanced Malignant Tumors.
Brief Title: First-in-Human Investigation of JMT108 Injection in Participants With Advanced Malignant Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shanghai JMT-Bio Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JMT108-001
Record Dates: First submitted 2025-03-06; First posted 2025-03-14 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2025-04

CONDITIONS: Advanced Malignant Tumors
MeSH Terms: interventions — pembrolizumab

STUDY DESIGN:
Intervention Model Description: This study is designed as an open-label, multi-center Phase 1 clinical study in participants with advanced malignant tumors to evaluate the safety, tolerability, PK characteristics, and preliminary anti-tumor activity of JMT108 injection, and to determine the RP2D/schedule for subsequent studies.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- JMT108 (Experimental)
  Interventions: Drug: JMT108; Drug: Pembrolizumab; Drug: Ivonescimab

INTERVENTIONS:
Drug: JMT108 — Intravenous (IV) administration every three weeks (D1) in a 3-week cycle.
Drug: Pembrolizumab — Intravenous (IV) administration every three weeks (D1) in a 3-week cycle.
Drug: Ivonescimab — Intravenous (IV) administration every three weeks (D1) in a 3-week cycle.

SUMMARY:
This study is designed as an open-label, multi-center Phase 1 clinical study in participants with advanced malignant tumors to evaluate the safety, tolerability, PK characteristics, and preliminary anti-tumor activity of JMT108 injection, and to determine the RP2D/schedule for subsequent studies.

ELIGIBILITY:
Inclusion Criteria:

1. Fully informed of the study, with good compliance and willing to provide written informed consent.
2. Male or female participants aged ≥18 years (at the time of obtaining informed consent).
3. Participants with histologically or cytologically confirmed advanced malignant tumors who are unresponsive or intolerant to all standard of care, or have no standard of care available. For locally advanced (stage IIIB/IIIC) or metastatic (stage IV) NSCLC without sensitive gene mutations, participants who have not received systemic treatment in the advanced stage and are unwilling to accept the current standard treatment can also be enrolled in the cohort expansion phase.
4. Participants with at least one evaluable tumor lesion in the Phase 1a dose-escalation phase; and at least one measurable lesion in the Phase 1a dose-expansion phase and Phase 1b (tumor lesions in the past radiation fields or that underwent locoregional therapy are generally not considered measurable lesions unless the lesion shows definite progression or persists three months after radiotherapy) according to RECIST v1.1.
5. Stage I: ECOG performance score ≤ 2. Stage II: ECOG performance score 0-1
6. Expected survival ≥ 3 months.
7. Adequate organ function status:

Hematology: PLT ≥ 100×109/L; Hb ≥ 90 g/L; ANC) ≥ 1.5×109/L (No blood transfusion, platelet transfusion, or hematopoietic stimulating factor therapy within 14 days prior to hematology test during the screening period); Liver function: AST and ALT ≤3×ULN (≤5×ULN if there is liver involvement by the tumor); TBIL ≤1.5×ULN; Renal function: Ccr > 50 ml/min (calculated by the Cockcroft-Gault formula); Coagulation function: APTT ≤ 1.5×ULN; INR ≤ 1.5×ULN; For participants on full - dose oral anticoagulant therapy, maintain a stable dosage for at least 14 days. If on warfarin, INR ≤ 3.0 with no active hemorrhage (e.g., no bleeding 14 days before the first dose of the investigational drug). Low molecular weight heparin use is permitted.

Albumin: ≥30 g/L (≥3.0 g/dL).

Exclusion Criteria:

1. Any other unapproved investigational drugs or treatments within 4 weeks prior to the first dose of the investigational drug (C1D1).
2. Chemotherapy, radiotherapy, biological therapy, endocrine therapy, targeted therapy, immunotherapy, or other anti-tumor therapies within 4 weeks prior to the first dose of the investigational drug, except in the following situations:

   Nitrosoureas or mitomycin C within 6 weeks prior to the first dose of the investigational drug; Use of oral fluoropyrimidines and small-molecule targeted drugs within 2 weeks or 5 half-lives of the drug (whichever is longer) prior to the first dose of the investigational drug; Use of herbal medicine/products with anti-tumor indications within 2 weeks prior to the first dose of the investigational drug.
3. Major surgery (excluding biopsy) or experienced severe trauma within 4 weeks prior to the first dose of the investigational drug, or plan to do major surgery during the study period.
4. Systemic corticosteroids or other immunosuppression therapy within 14 days prior to the first dose of the investigational drug. Except for the following situations: use of physiological replacement doses of hydrocortisone or other equivalent doses of hormones (i.e., prednisone ≤10 mg/day or other equivalent doses of hormones); use of topical, ocular, intra-articular, intranasal, and inhaled corticosteroid therapy; use of short-course glucocorticoids for prophylaxis (e.g., prevention of contrast allergy).
5. Live vaccines within 4 weeks prior to the first dose of investigational drug. Note: Seasonal influenza vaccines are inactivated vaccines in a broad sense and are allowed. Intranasal influenza vaccines are live vaccines and are not permitted.
6. History of hematopoietic stem cell transplant or organ transplant.
7. AEs from prior therapy which have not recovered to Grade ≤1 or baseline as per NCI CTCAE v5.0 (excluding toxicities evaluated by the investigator to have no safety risk, such as alopecia, Grade 2 peripheral neurotoxicity, hypothyroidism stabilized with hormone replacement therapy, etc.).
8. Active central nervous system metastases and/or leptomeningeal metastases. Participants with brain metastases who have confirmed progression-free status by imaging examinations for at least 4 weeks after treatment and who have not required hormonal or antiepileptic therapy for at least 2 weeks may be considered for enrollment.
9. History of interstitial lung disease or pneumonitis.
10. History of serious cardiovascular and cerebrovascular diseases.
11. Active or recurrent autoimmune diseases (such as systemic lupus erythematosus, arthritis, vasculitis, etc.).
12. History of Grade ≥3 immune-related AE or Grade ≥2 immune-related myocarditis considered related to prior immune modulatory therapytherapy.
13. Hemorrhage of Grade ≥2 as per NCI CTCAE v5.0 within 4 weeks prior to the first dose of the investigational drug.

    -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 436 (Estimated)
Dates: Start 2025-04-11 (Actual); Primary Completion 2028-03-30 (Estimated); Study Completion 2029-03-30 (Estimated)

PRIMARY OUTCOMES:
Dose-Limiting Toxicity(DLT) | Approximately 28 days.
  To evaluate the safery of JMT108 in subjects.
Adverse Events (AEs) | through study completion, an average of 1 year
  To evaluate the safery of JMT108 in subjects

SECONDARY OUTCOMES:
Maximum plasma concentration (Cmax) | through study completion, an average of 1 year
  To evaluate the systemic pharmacokinetics of JMT108 in subjects.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality, China